CLINICAL TRIAL: NCT05757323
Title: A Randomized, Controlled, Double-blind Parallel Group Trial to Study the Effects of an Infant Formula Containing Partially Hydrolysed Proteins on Growth and Tolerance in Healthy Term Infants
Brief Title: The Effects of an Infant Formula Containing Hydrolysed Proteins on Growth and Tolerance in Healthy Term Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FrieslandCampina (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HerA
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Growth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- test formula (Experimental): hydrolysed protein-based infant formula
  Interventions: Other: infant formula based on hydrolyzed protein
- control formula (Active Comparator): standard intact protein-based formula
  Interventions: Other: infant formula based on intact protein

INTERVENTIONS:
Other: infant formula based on hydrolyzed protein — infant formula based on hydrolysed protein
  Arms: test formula
Other: infant formula based on intact protein — infant formula based on intact protein
  Arms: control formula

SUMMARY:
In this clinical trial, weight gain (primary objective), and additional anthropometry (secondary objectives), of infants exclusively consuming a hydrolysed protein-based infant formula were evaluated and compared to a standard intact protein-based formula over a period of at least three months, until the age of 17 weeks.

DETAILED DESCRIPTION:
In this clinical trial, weight gain (primary objective), and additional anthropometry (secondary objectives), of infants exclusively consuming a hydrolysed protein-based infant formula were evaluated and compared to a standard intact protein-based formula over a period of at least three months, at the age of 8, 13, and 17 weeks. 345 healthy term infants, exclusively formula-fed were included.

ELIGIBILITY:
Inclusion criteria:

* Full-term infants (born at gestational age =37 weeks).
* Healthy birthweight (according to WHO Child Growth Standards): between 2500 and 4200 g, retrieved from medical records
* Boys and girls
* Apparently healthy at birth and screening
* Weight-for-age Z-score (WAZ), weight-for-length (WHZ), and length-for-age (LAZ) Z-scores at screening within the normal range according to WHO Child Growth Standards (i.e. -2 = WAZ,WHZ,LAZ = 2)
* Age at enrolment: =28 days of age
* Exclusively formula fed for at least 5 days prior to inclusion
* Exclusively formula fed during the entire intervention period
* Parents agreeing to initiate complementary feeding after finalization of the study
* Being available for follow up until the age of approximately 3.5 months
* Written informed consent from parent(s) and/or legal guardian(s) aged =18 years

Exclusion criteria:

* Gestational age <37 weeks
* Birth weight <2500 g or >4200 g
* Age at enrolment: >28 days
* Severe acquired or congenital diseases, mental or physical disorders, including cow's milk protein allergy, lactose intolerance and diagnosed medical conditions that are known to affect growth (i.e. GI disorders)
* Illness at screening/inclusion
* Incapability of parents to comply with the study protocol
* Illiterate parents (i.e. not able to read and write in local language)
* Participation in another clinical trial
* Unwillingness to accept the formula supplied by the study as the only formula for their child during study participation
* infants fed a special diet other than standard, non-hydrolysed, cow's or goat's milk based infant formula

Ages: 5 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 345 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
weight gain | until 17 weeks of age
  weight gain in g/day

SECONDARY OUTCOMES:
Weight | until 17 weeks of age
  Weight in g
Length | until 17 weeks of age
  length in cm
head circumference | until 17 weeks of age
  head circumference in cm
BMI | until 17 weeks of age
  BMI in kg/m2
WAZ | until 17 weeks of age
  weight-for-age Z-score
LAZ | until 17 weeks of age
  length-for-age Z-score
WHZ | until 17 weeks of age
  weight-for-height Z-score
BMI-for-age Z-score | until 17 weeks of age
  BMI-for-age Z-score
head circumference-for-age Z-score | until 17 weeks of age
  head circumference-for-age Z-score

OTHER OUTCOMES:
formula intake | until 17 weeks of age
  formula intake in ml

CONTACTS AND LOCATIONS:
Overall Officials: Yannis Manios, Prof, Principal Investigator — Harokopio University
Locations (3):
- Greece (3):
  - Department of Nutrition and Dietetics, University of Thessaly, Trikala, Thessaly
  - Harokopio University, Athens
  - Department of Nutritional Sciences, International Hellenic University, Thessaloniki

REFERENCES:
- [Derived] Kantaras P, Kokkinopoulou A, Hageman JHJ, Hassapidou M, Androutsos O, Kanaki M, Bovee-Oudenhoven I, Karaglani E, Kontochristopoulou AM, Bos R, Manios Y. Growth and gut comfort of healthy term infants exclusively fed with a partially hydrolysed protein-based infant formula: a randomized controlled double-blind trial. Front Pediatr. 2024 May 17;12:1328709. doi: 10.3389/fped.2024.1328709. eCollection 2024. PMID 38827219
- See also: first registration of the trial (register is closed, so not able to enter new data) — https://trialsearch.who.int/Trial2.aspx?TrialID=NL9536